CLINICAL TRIAL: NCT02650648
Title: Phase I Study of the Humanized Anti-GD2 Antibody Hu3F8 and Allogeneic Natural Killer Cells for High-Risk Neuroblastoma
Brief Title: Humanized Anti-GD2 Antibody Hu3F8 and Allogeneic Natural Killer Cells for High-Risk Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-272; 5415 (Other: OPD grant number)
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma; High-Risk
Keywords: Humanized Anti-GD2 Antibody Hu3F8; Allogeneic Natural Killer Cells; rIL-2; 15-272
MeSH Terms: conditions — Neuroblastoma | interventions — Cyclophosphamide; naxitamab

ARMS (1):
- Humanized Anti-GD2 Antibody Hu3F8 (Experimental): This is a phase I study to assess the safety and feasibility of combining HLA-mismatched (KIR ligand incompatible) NK cells with hu3F8 in high-risk NB patients. Following chemotherapy, patients will be treated in sequential groups with a minimum of 3 patients/ dose of NK cells. Three dose levels of NK cells, starting at dose level 1, will be evaluated in this treatment protocol. The goal dose for each dose level is the high boundary (e.g. 9.9x10^6/kg in level 1; 14.9x10^6/kg in level 2, etc), but a range is provided to allow for cases where the goal dose cannot be achieved.
  Interventions: Drug: cyclophosphamide; Biological: NK cells; Biological: hu3F8; Drug: rIL-2

INTERVENTIONS:
Drug: cyclophosphamide — chemotherapy with intravenous (IV) cyclophosphamide 50mg/kg/day (for patients with body weight<70kg) or 1500mg/m^2/day (for patients with body weight ≥70kg) for two days (days -6 and -5).
  Other Names: Cytoxan®
Biological: NK cells — Day 0: NK cell infusion. NK cells are resuspended in Normasol at a concentration no less than 5 x 10^6cells/mL. The patient is pre-medicated as per standard cell product infusion. The cell product is infused through a central venous catheter. Patients will be evaluated clinically by vital signs pre- and approximately 30 minutes post infusion of NK cells and thereafter at approximately 1 hour intervals for 4 hours.
Biological: hu3F8 — On Days -1, +1, +5, +7 and +9 hu3F8 is administered at 1.68 mg/kg/day and infused over ~30-90 minutes
Drug: rIL-2 — On day 0, daily from +2 through +4, day +6, and day +8, rIL-2 is administered subcutaneously at 6 x 10^5 U/m^2/day.

SUMMARY:
This is a phase I study. The purpose of this study is to see if it is safe and feasible to give the participant cyclophosphamide (a type of chemotherapy), natural killer (NK) cells, and an antibody called Hu3F8 as a treatment for neuroblastoma. NK cells are a type of white blood cell.

Funding Source- FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by international criteria,.e., histopathology (confirmed by the MSKCC Department of Pathology) or bone marrow metastases plus high urine catecholamine levels.
* High-risk NB as defined by risk-related treatment guidelines1 and the International NB Staging System, i.e., stage 4 with (any age) or without (>365 days of age) MYCN amplification, MYCN-amplified stage 3 (unresectable; any age), or MYCN-amplified stage 4S.
* Patients must have a history of tumor progression or persistent disease or failure to achieve complete response following standard therapy.
* Patients must have evaluable (microscopic marrow metastasis, elevated tumor markers, positive MIBG or PET scans) or measurable (CT, MRI) disease documented after completion of prior systemic therapy.
* Disease staging approximately within one month of treatment
* Prior treatment with murine and hu3F8 is allowed. Patients with prior m3F8, hu3F8, ch14.18 or hu14.18 treatment must have a negative HAHA antibody titer. Human anti-mouse antibody (HAMA) positivity is allowed.
* Eligible NK donor
* Children and adults are eligible
* Signed informed consent indicating awareness of the investigational nature of this program.

Donor Inclusion Criteria

* Donor is blood-related and HLA-haploidentical to the recipient.
* Donor has undergone serologic testing for transmissible diseases as per blood banking guidelines for organ and tissue donors. Tests include but are not limited to: Hepatitis B Surface Antigen, Hepatitis B Surface Antibody, Hepatitis B Core Antibody, Hepatitis C antibody, Epstein-Barr Virus Antibody, HIV, HTLV I and II, Varicella Zoster (Herpes Zoster), Herpes Simplex Antibody, Cytomegalovirus Antibodies, Syphilis (RPR profile) for adolescents and adults, measles for pediatric patients, West Nile Virus, Chagas screen, and Toxoplasma antibodies. Donor must have normal negative test results for HIV, HTLV I and II, and West Nile Virus. Donor exposure to other viral pathogens will be discussed on a case-by-case basis by investigators.
* Donor must be able to undergo leukopheresis for total volume of 10-15 liters.
* There is no age restriction for the donor.

Exclusion Criteria:

* Patients with CR/VGPR disease
* Existing severe major organ dysfunction, i.e., renal, cardiac, hepatic, neurologic, pulmonary, or gastrointestinal toxicity > grade 3 except for hearing loss, alopecia, anorexia, nausea, hyperbilirubinemia and hypomagnesemia from TPN, which may be grade 3
* ANC should be >500/uL
* Platelet count >75K/uL.
* History of allergy to mouse proteins
* Active life-threatening infection
* Inability to comply with protocol requirements
* Women who are pregnant or breast-feeding

Donor Exclusion Criteria:

* Cardiac risk factors precluding ability to undergo leukopheresis
* Concurrent malignancy or autoimmune disease
* Donor is pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
The number patient responses observed at each dose level | 2 years
  as defined by International NB Response Criteria. Disease status is defined by the International NB Response Criteria. Complete response/remission (CR): no evidence of disease. Very good partial response/remission (VGPR): >90% decrease in all disease parameters, except bone scan unchanged or improved; bone marrow must be free of disease. Partial response/remission: >50% decrease in all disease parameters, except bone scan unchanged or improved; no more than 1 positive bone marrow site. Mixed response: >50% decrease in >1 but not all disease markers. Stable disease: <50% decrease in all tumor markers. Progressive disease: new lesion, or >25 % increase in any disease marker.

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel Modak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/